CLINICAL TRIAL: NCT00383071
Title: A Phase II Vaccine Dose Finding Pilot Study for Development of an Anti-Influenza A (H5N1) Intravenous Hyper-Immune Globulin
Brief Title: Development of Immune Globulin Treatment for Avian Flu
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Cannot get enough plasma to manufacture IVIG for human trials
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 06-I-0235; 060235 (Other: NIH Protocol Services)
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2016-04

CONDITIONS: Infectious Diseases; Influenza; Avian Flu
Keywords: Apheresis; Avian Flu; Healthy Volunteers; Infectious Diseases; IVIG; Healthy Volunteer; HV
MeSH Terms: conditions — Communicable Diseases; Influenza, Human; Influenza in Birds | interventions — Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Active Comparator): H5N1 vaccine - 90 mcg IM every 4 week x 4 doses Apheresis - if HAI titer above 1:160
  Interventions: Biological: H5N1 vaccine; Procedure: Apheresis
- Cohort 2 (Active Comparator): H5N1 vaccine - 120 mcg IM every 4 week x 4 doses Apheresis - if HAI titer above 1:160
  Interventions: Biological: H5N1 vaccine; Procedure: Apheresis
- Cohort 3 (Active Comparator): H5N1 vaccine - 180 mcg IM every 4 week x 4 doses Apheresis - if HAI titer above 1:160
  Interventions: Biological: H5N1 vaccine; Procedure: Apheresis
- Cohort 4 (Active Comparator): H5N1 vaccine - 180 mcg IM every 4 weeks x 2 doses, injection site randomized to either deltoid or gluteus Apheresis - if HAI titer above 1:160
  Interventions: Biological: H5N1 vaccine; Procedure: Apheresis

INTERVENTIONS:
Biological: H5N1 vaccine — Monovalent subvirion H5N1 vaccine (rgA/Vietnam/1203/2004) 90 mcg/mL Manufactured by Sanofi Pasteur Inc, Swiftwater, PA.
Procedure: Apheresis — Once subjects achieved a high antibody titer (>1:160), they could begin apheresis to collect plasma.

SUMMARY:
This study will determine how best to use a vaccine for generating high levels of antibodies called immune globulins (IVIG) in people, which, in turn, can be collected and used to develop a possible treatment for avian influenza (bird flu). Immune globulins are proteins made by the body that attack the influenza virus. This study will use an experimental bird flu vaccine to stimulate immune globulin production in healthy people. The vaccine is similar to the regular influenza vaccine and has been studied in more than 450 people. This study will use high doses of the vaccine to generate high antibody levels that can be collected for producing the new treatment.

Healthy adults between 18 and 60 years of age who weigh at least 110 pounds may be eligible for this study. Candidates are screened with a medical history and physical examination.

Participants are given one of three doses of the vaccine, depending on when they enter the study. The first 25 people enrolled receive a dose of 90 micrograms (mcg). If this dose is well tolerated, the next 25 people receive 120 mcg, and if this dose is also well tolerated, the last 25 people receive 180 mcg. Vaccination consists of either two shots (one in the muscle of each arm) or one shot in the buttock on four occasions. Subjects are vaccinated on four occasions, each 4 weeks apart. On the day of each vaccination, subjects provide a blood sample to evaluate blood counts, chemistries, and antibody levels, and to test for HIV, hepatitis B and C, syphilis, and antibody against avian flu. For 7 days after each vaccination, subjects keep a diary card to record any symptoms, such as pain, fever, muscle aches, or others. At the end of the 7 days, they are contacted by study staff to report the symptoms.

In addition to the vaccinations, subjects undergo apheresis to collect IVIG once their blood test shows moderately high antibody levels. For this procedure, blood is collected through a needle in an arm vein and flows through a catheter (plastic tube) into a machine that separates the blood cells from the antibodies and protein. The antibodies and protein are collected and the rest of the blood is returned to the body. Subjects are asked to undergo at least three apheresis procedures.

...

DETAILED DESCRIPTION:
Avian influenza presents a threat of a future pandemic. Over 200 people have been infected with the influenza A H5N1 virus, and the mortality is near 60 percent. Optimal therapy is not known, and failures of and resistance to currently available anti-virals have been reported.

The primary purpose of this Protocol is to determine the optimal vaccination schedule that creates a pool of hyper immunized individuals with high titer anti-influenza A (H5N1) antibodies. The Protocol will consist of a dose escalation study to determine the optimal vaccination dose and number of vaccinations. There are stopping rules based on the number and severity of adverse events that occur between the doses and between the cohorts. The optimal vaccination schedule that is determined could then be used in a larger population to develop a high titer anti-influenza A (H5N1) intravenous hyper-immune globulin (IVIG).

After all vaccinations have occured, and if an adequate antibody titer is reached in this study population, subjects will begin apheresis. Each subject will be asked to participate in 3 apheresis sessions, but may participate in up to 10 apheresis sessions.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years old, and < 60 years old.
2. Adequate clinical parameters (all of the following):

   * Afebrile (temperature < 38° C)
   * Systolic blood pressure >100 & <180 mmHg
   * Diastolic blood pressure >50 & <100 mmHg
   * Heart rate between 40-100 beats/minute
3. Weight ≥ 110 pounds (50kg)
4. Adequate peripheral venous access for plasmapheresis (as judged by the examiner)
5. Females of child-bearing potential must (one of the following):

   * Be surgically sterile.
   * Be abstinent (or willing to be) 4 weeks prior to date of screening evaluation through the last apheresis session (estimate 6 months).
   * Use oral contraceptives, or other form of hormonal birth control including hormonal vaginal rings or transdermal patches, and have been using these for 3 months prior to date of screening evaluation through the last apheresis session (estimate 6 months).
   * Use an intra-uterine device (IUD) as birth control 4 weeks prior to date of screening evaluation through the last apheresis session (estimate 6 months).
   * Use (by ensuring her male partner(s) uses) barrier contraception (condom) with a spermicide as birth control 4 weeks prior to date of screening evaluation through the last apheresis session (estimate 6 months).

Exclusion Criteria:

1. Has a medical history of

   * Thrombocytopenia or other blood dyscrasias
   * congestive heart failure
   * pulmonary hypertension
   * bleeding diathesis or therapeutic anticoagulation
   * HIV/AIDS
   * Hepatitis B
   * Hepatitis C
   * Known history of hepatitis after the 11th birthday.
   * Trypanosomiasis (Chagas' disease and sleeping sickness)
   * Leishmaniasis (Kala-azar)
   * Filariasis
   * Q fever
   * Yaws
   * Allergy to eggs, thimerosal, or other components of the vaccine
   * Severe reactions following immunization with contemporary influenza virus vaccines
   * Autoimmune disease or a history of Guillain-Barré
2. History of cancer that meets any one of the following criteria:

   * Non-melanoma skin cancers within the last 1 year
   * Melanoma or any other cancer (excluding non-melanoma skin cancers) at any time
3. Medication history that includes any of the following:

   * Current use of oral or parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs
   * Finasteride (Proscar, Propecia) within the last 1 month.
   * Isotretinoin (Accutane) within the last 1 month.
   * Acitretin (Soriatane) within the last 3 years.
   * Etretinate (Tegison) at any time.
   * Dutasteride (Avodart) within the last 6 months.
   * Growth hormone made from human pituitary glands at any time.
   * Beef insulin from the United Kingdom at any time.
4. Has ever had any of the following:

   * Sexual contact with someone known to have HIV.
   * Had a relative with Creutzfeldt-Jakob Disease, or been told that this disease is inherited within the family.
   * Received blood transfusion in the United Kingdom.
   * History of receiving money, drugs or other payment for sex.
   * History of receiving clotting factor concentrates.
   * History of a dura mater graft.
   * History of babesiosis.
   * For male donors, history of sexual contact with another male.
   * Used needles to take drugs, steroids, or other medications not prescribed by a physician.
   * Was born, lived in, had blood donation in or ever had sexual contact with anyone who lived in Cameroon, Central African Republic, Chad, Congo, Equatorial Guinea, Gabon, Niger, or Nigeria after 1977.
   * History of living 3 or more months total (need not be consecutive) in the UK from 1980-1996.
   * History of living 5 or more years total (need not be consecutive) in Europe since 1980.
   * History of living 6 or more months total (need not be consecutive) on a U.S. military base in Europe from 1980-1996 (specifically from 1980 through 1990 in Belgium, the Netherlands, or Germany, and from 1980 through 1996 in Spain, Portugal, Turkey, Italy or Greece).
5. Within the last 3 weeks received the seasonal (conventional trivalent) flu vaccine
6. Within the last 8 weeks:

   • Was vaccinated with the small pox vaccine, or was in close contact with someone who was vaccinated (i.e., close family member).
7. Within the last 3 months has:

   • Current or previous participation in any other apheresis procedures/protocols (not related to this protocol).
8. Within the last 4 months has had:

   • A blood donation of a double unit of red cells.
9. Within the last 12 months has:

   * Received any blood or blood component.
   * Donated blood at a paid donation center (donations at a hospital blood bank do not apply).
   * History of unsafe (multiple-use equipment) tattoo, acupuncture, or piercing practices.
   * Received an organ transplant.
   * Received a bone or skin graft.
   * Lived with someone who has any type of hepatitis.
   * Traveled to areas with malaria.
   * Been incarcerated for more than 72 hours.
   * Oral or inhalation use of illegal drugs (i.e. those not prescribed by a physician).
   * Had or has been treated (with or without confirmatory diagnosis) for syphilis or gonorrhea
10. Within the last 12 months has had sexual contact with (any of the following):

    * An individual having viral hepatitis.
    * A prostitute or anyone else who takes money or drugs or other payment for sex.
    * Anyone who has ever used needles to take drugs, steroids, or anything else not prescribed by their doctor.
    * Anyone who has hemophilia or has used clotting factor concentrates.
    * For females, a male who has ever had sexual contact with another male.
11. Participation in medical research that includes:

    * Protocols that are currently ongoing or will start during the duration of this study that require more than 100cc of blood to be given in any 6-week period of time.
    * Administration of any unlicensed drug within the last 3 months or during the duration of this study.
    * Administration of any unlicensed vaccine within the last 12 months or during the duration of this study.
12. Currently pregnant (if known).
13. Any condition that, in the opinion of the investigator, would render vaccination unsafe, would interfere with the antibody response or the evaluation of these responses, or would place the subject at increased risk of injury from apheresis.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2006-08; Primary Completion 2010-03 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Clifford Lane, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Morse SS. Factors in the emergence of infectious diseases. Emerg Infect Dis. 1995 Jan-Mar;1(1):7-15. doi: 10.3201/eid0101.950102. PMID 8903148
- [Background] de Jong MD, Tran TT, Truong HK, Vo MH, Smith GJ, Nguyen VC, Bach VC, Phan TQ, Do QH, Guan Y, Peiris JS, Tran TH, Farrar J. Oseltamivir resistance during treatment of influenza A (H5N1) infection. N Engl J Med. 2005 Dec 22;353(25):2667-72. doi: 10.1056/NEJMoa054512. PMID 16371632
- [Background] Chotpitayasunondh T, Ungchusak K, Hanshaoworakul W, Chunsuthiwat S, Sawanpanyalert P, Kijphati R, Lochindarat S, Srisan P, Suwan P, Osotthanakorn Y, Anantasetagoon T, Kanjanawasri S, Tanupattarachai S, Weerakul J, Chaiwirattana R, Maneerattanaporn M, Poolsavathitikool R, Chokephaibulkit K, Apisarnthanarak A, Dowell SF. Human disease from influenza A (H5N1), Thailand, 2004. Emerg Infect Dis. 2005 Feb;11(2):201-9. doi: 10.3201/eid1102.041061. PMID 15752436
- [Derived] Lu H, Khurana S, Verma N, Manischewitz J, King L, Beigel JH, Golding H. A rapid Flp-In system for expression of secreted H5N1 influenza hemagglutinin vaccine immunogen in mammalian cells. PLoS One. 2011 Feb 28;6(2):e17297. doi: 10.1371/journal.pone.0017297. PMID 21386997
- [Derived] Beigel JH, Voell J, Huang CY, Burbelo PD, Lane HC. Safety and immunogenicity of multiple and higher doses of an inactivated influenza A/H5N1 vaccine. J Infect Dis. 2009 Aug 15;200(4):501-9. doi: 10.1086/599992. PMID 19569973
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-I-0235.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2: 120 mcg: 120 mcg every 28 days x 4 doses. Subjects chose vaccination in arm or buttock.
- Cohort 3: 180 mcg; Cohort 1: 90 mcg: 180 mcg every 28 days x 4 doses. Subjects chose vaccination in arm or buttock.
- Cohort 4: 180 mcg: 120 mcg every 28 days x 2 doses. Subjects randomized to receive vaccination in arm or buttock.
Period: Overall Study
Arm/Group | Cohort 2: 120 mcg | Cohort 3: 180 mcg | Cohort 4: 180 mcg | Cohort 1: 90 mcg
Started | 25 | 25 | 51 | 25
Completed | 25 | 21 | 44 | 22
Not Completed | 0 | 4 | 7 | 3

BASELINE CHARACTERISTICS:
Population: All subjects enrolled into the study
Groups:
- 120 mcg: 120 mcg IM every 4 weeks for 4 vaccinations
- 180 mcg: 180 mcg IM every 4 weeks for 4 vaccinations
- 180 mcg Cohort 4: 180 mcg IM every 4 weeks for 2 vaccinations
- 90 mcg: 90 mcg IM every 4 weeks for 4 vaccinations
- Total: Total of all reporting groups
Arm/Group | 120 mcg | 180 mcg | 180 mcg Cohort 4 | 90 mcg | Total
Number analyzed (Participants) | 25 | 25 | 51 | 25 | 126
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 1 | 0 | 0 | 0 | 1
  BTWN | 24 | 25 | 51 | 25 | 125
  GTE65 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 20 | 15 | 60
  Male | 13 | 12 | 31 | 10 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic | 2 | 0 | 5 | 0 | 7
  Not Hispanic or Latino | 23 | 25 | 46 | 24 | 118
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 1 | 1 | 6
  Hawaiian | 0 | 0 | 0 | 0 | 0
  Black | 2 | 6 | 8 | 5 | 21
  White | 19 | 15 | 40 | 17 | 91
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 3 | 0 | 2 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Safety of H5N1 Vaccine as Measured by Adverse Events
Description: The number of subjects experiencing adverse events after receiving H5N1 vaccine
Time Frame: Day 28, 56, 84
Population: Primary outcome measure was safety, so below listed numbers are safety population used in AE list.
Measure: Number; unit: participants
Groups:
- 180 mcg Cohort 4: 120 mcg IM every 4 weeks for 2 vaccinations
Arm/Group | 90 mcg | 120 mcg | 180 mcg | 180 mcg Cohort 4
Number analyzed (Participants) | 25 | 25 | 25 | 51
participants | 24 | 24 | 25 | 46

ADVERSE EVENTS:
Groups:
- 120 mcg: 120 mcg every 28 days x 4 doses
- 180 mcg: 180 mcg every 28 days x 4 doses
- 180 mcg Cohort 4: 180 mcg every 28 days x 2 doses
- 90 mcg: 90 mcg every 28 days x 4 doses
Arm/Group | 120 mcg | 180 mcg | 180 mcg Cohort 4 | 90 mcg
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25 | 2/51 | 1/25
Other Adverse Events (participants affected / at risk) | 24/25 | 25/25 | 46/51 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 120 mcg (N=25) | 180 mcg (N=25) | 180 mcg Cohort 4 (N=51) | 90 mcg (N=25)
Sickle-cell Disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Idiopathic thrombocytopenia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 120 mcg (N=25) | 180 mcg (N=25) | 180 mcg Cohort 4 (N=51) | 90 mcg (N=25)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis, external ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis, middle ear (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal gas pains (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 4 (4) | 3 (3)
Oral aphthous ulcer(s) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste changes (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute pain (General disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1)
Erythema at injection site (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 5 (5) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Influenza-like disease (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Reaction (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Injection site tenderness (General disorders) | 17 (17) | 20 (20) | 32 (32) | 20 (20)
Malaise (General disorders) | 8 (8) | 6 (6) | 10 (10) | 6 (6)
Pain at injection site (General disorders) | 11 (11) | 12 (12) | 20 (20) | 16 (16)
Pruritis associated with injection (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Swelling at injection site (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adhesions, small bowel (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abnormal serum CPK (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased hemoglobin (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Decreased serum albumin (Investigations) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Elevated ALT(SGPT) (Investigations) | 2 (2) | 1 (1) | 1 (1) | 5 (5)
Elevated AST(SGOT) (Investigations) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Elevated blood pressure reading without diagnosis of hypertension (Investigations) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Elevated Hematocrit (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated Hemoglobin (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated serum bilirubin (Investigations) | 9 (9) | 8 (8) | 19 (19) | 6 (6)
Elevated serum creatinine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated Uric Acid (hyperuricemia) (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Heart murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Investigations) | 8 (8) | 2 (2) | 6 (6) | 2 (2)
Hyperkalemia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatremia (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypophosphatemia (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Platelets, decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - other (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Backache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bone fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis of hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fasciculations (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5) | 8 (8) | 6 (6)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (TMJ) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alterations in neuro-sensory functioning (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance of skin sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 12 (12) | 8 (8) | 13 (13) | 10 (10)
Light headedness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasovagal episode (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sleep Disturbance (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (UTI) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atypical squamous cell of undetermined significance (ASCUS) (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hypertrophy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2)
Allergic rhinitis (nonseasonal) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (seasonal) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Common cold (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nonspecific rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (3) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Idiopathic thrombocytopenia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elective surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 4 (4) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes